CLINICAL TRIAL: NCT00441389
Title: Infectious Etiology of Acute Exacerbations of COPD in Hong Kong
Brief Title: Infectious Etiology of Acute Exacerbations of COPD
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Other Study IDs: Resp/ko/2006/003
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Bacteria; Viruses; COPD; infectious etiology for acute exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Virus Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the infectious etiology related to acute exacerbation of COPD in Hong Kong

DETAILED DESCRIPTION:
Subject recruitment

Patients admitted with AECOPD will be recruited for this study. AECOPD is defined a patient with background COPD with at least two of the major symptoms (increased dyspnoea, increased sputum purulence, increased sputum amount) or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, cough) for at least two consecutive days. Informed written consent will be obtained. Exclusion criteria included patients with myocardial infarction within the preceding 6 months, unstable angina, congestive heart failure (with New York Heart Association class III or IV) and those who cannot give consent for the study.

Demographic data and management in hospital Detailed information on the COPD exacerbations including demographic data (age, sex, height and weight, background illness and functional status), symptoms, blood test results and length of hospital stay will be recorded. In addition, chest radiographs will be assessed by the investigators (respiratory physicians) and abnormalities like pneumonic changes will be noted. The type and duration of antibiotics used will be recorded. Any non-invasive ventilation used or intensive care unit admissions will be assessed.

Microbiological test Routine and mycobacterial sputum culture, nasopharyngeal aspirate for viruses, blood for atypical pneumonia serology and urine for pneumococcal and legionella species will be collected and processed by standard microbiological techniques in the microbiology laboratory of the Prince of Wales Hospital for each patient upon admission to medical wards. Convalescent atypical pneumonia serology will be collected 14 days later. The sensitivity of the cultured organisms to antibiotics will also be assessed.

Follow up of progress of patients post discharge During follow up, lung function (including spirmotery pre and post bronchodilator and 6 minutes walk test) of the patient will be monitored at 1 month post discharge and subsequently at 6 months interval. The degree of dyspnoea will be assessed by modified Medical Research Council dyspnoea scale (MMRC) and quality of life will be assessed by St George's Respiratory Questionnaire (SGRQ) at 1 month and 12 months post discharge. Patients will be followed up in the lung function laboratory for 2 year (at 1 month, 6 months, 12 months, 18 months and 24 months). The patient and the family will be contacted if the patient failed to return for appointments. Death from any cause and from special respiratory causes will be recorded. Cause of death will be reviewed by the investigators by reviewing the medical record and death certificate.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with AECOPD will be recruited for this study.
* AECOPD is defined a patient with background COPD16 with at least two of the major symptoms (increased dyspnoea, increased sputum purulence, increased sputum amount) or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, cough) for at least two consecutive days.
* Informed written consent will be obtained.

Exclusion Criteria:

* Exclusion criteria included patients with myocardial infarction within the preceding 6 months, unstable angina, congestive heart failure (with New York Heart Association class III or IV) and those who cannot give consent for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-05; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Fanny KO, FCCP, Principal Investigator — Chinese University of Hong Kong